CLINICAL TRIAL: NCT07103564
Title: The Evaluation of the Effect of Local Melatonin Application Around Immediately Placed Implants in the Maxillary Premolars (Randomized Controlled Clinical Trial)
Brief Title: The Effect of Local Melatonin Application Around Immediately Placed Implants in the Maxillary Premolar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Lecturer of Dental Public Health and biostatistical consultanat, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0812-12/2023
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Dental Implants; Osteoprotegerin; Melatonin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- melatonin therapy (Experimental)
  Interventions: Other: Immediately placed implant in maxillary premolars with local melatonin application
- No melatonin (Active Comparator)
  Interventions: Other: Immediately placed implant in maxillary premolars without local melatonin application

INTERVENTIONS:
Other: Immediately placed implant in maxillary premolars with local melatonin application — Patients will receive immediately placed implants with local melatonin powder (3mg) application.
  Arms: melatonin therapy
Other: Immediately placed implant in maxillary premolars without local melatonin application — Patients will receive immediately placed implants without local melatonin application.
  Arms: No melatonin

SUMMARY:
Background: Immediate implants provide ideal three-dimensional positioning compared to conventional implants. There may be a gap between the surface of the implant and the bone walls of the socket when it is inserted into a recently extracted alveolus. To compensate for this, various grafting materials are used. Recently, melatonin has gained significant attention because of its inhibitory action on bone resorption through upregulating the expression of osteoprotegerin, which acts as a decoy receptor for RANKL and inhibits its binding to osteoclast precursors thereby inhibiting osteoclast formation and activity. So, we will conduct this study to evaluate the effects of local melatonin application around immediately placed implants.

Aim of the study: To evaluate the effectiveness of adding local melatonin around immediately placed implants in maxillary premolars.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-restorable maxillary premolars with sufficient bone quantity to receive the dental implant without the need for bone graft.
* Patients with no local or systemic pathology that can interfere with normal wound healing.
* Non-smokers.
* Patients who are properly motivated to complete follow-up visits

Exclusion Criteria:

* Patients with uncontrolled medical conditions that can affect surgical outcome or bone and wound healing. (ex: uncontrolled diabetes mellitus)
* Patients with periapical pathology that may contraindicate immediate implant placement.
* History of receiving irradiation in the head and neck region

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Change in Osteoprotegerin | Baseline, 1 month, and 3 months
  OPG (Ng/ml) level will be measured preoperatively, 1 and 3 months post operatively, to evaluate the bone healing activity. The level will be evaluated by collecting 5 ml of peripheral blood in blank tubes and will be allowed for complete clotting and will be centrifuged at 1000 g for 15 min. The separated serum will be then stored at -20 0C.
Change in bone volume | Baseline and 6 months
  CBCT scans will be obtained to measure change in bone volume
Change in bone level | Baseline and 6 months
  CBCT scans will be obtained to measure change in bone level
Change in bone density | Baseline and 6 months
  CBCT scans will be obtained to measure change in bone density

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Alexandria University, Alexandria, Egypt